CLINICAL TRIAL: NCT02793349
Title: ABSORB BTK Study: A Prospective, Multi-center, Controlled Clinical Evaluation of the Use of a Bioresorbable Drug Eluting Stent (Absorb, Abbott Vascular) in the Arterial Vasculature Below the Knee
Brief Title: The ABSORB Bioresorbable Scaffold Below the Knee (BTK) Study
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Company have withdrawn the product
Sponsor: The University of New South Wales (Other)
Responsible Party: Principal Investigator, Ramon Varcoe, Principal Investigator, The University of New South Wales
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HREC 15/051
Record Dates: First submitted 2016-06-03; First posted 2016-06-08 (Estimated); Last update posted 2019-04-17 (Actual); Status verified 2019-04

CONDITIONS: Ischemia; Peripheral Arterial Disease (PTA; Arterial Occlusive Diseases
Keywords: angioplasty; stents; polymers; absorbable implants
MeSH Terms: conditions — Ischemia; Peripheral Arterial Disease; Truncus Arteriosus, Persistent; Arterial Occlusive Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Bioresorbable Vascular Scaffold (Experimental): Absorb Bioresorbable Vascular Scaffold
  Interventions: Device: Absorb Bioresorbable Vascular Scaffold

INTERVENTIONS:
Device: Absorb Bioresorbable Vascular Scaffold — Absorb Bioresorbable Vascular Scaffold
  Other Names: BVS

SUMMARY:
ABSORB BTK Study: A prospective, multicenter, controlled clinical evaluation of the use of a bioresorbable drug eluting stent in the arterial vasculature below the knee

DETAILED DESCRIPTION:
The aim of this study is to evaluate the performance of a bioresorbable vascular scaffold (BVS) coated with the drug Everolimus. This will be used to treat short length blockages of up to 55mm (5.5cm) in arteries below the knee.

This will be performed to treat patients who have severe leg pain or have developed skin ulcers or gangrene which are not healing due to insufficent blood supply. The ABSORB Everolimus Eluting Bioresorbable Vascular Scaffold works on similar principles of drug eluting stents which have been used for a considerable time in treating blocked arteries. However this product consists of a scaffold coated with a drug so rather than leaving a metallic stent in the blood vessel, this product primarily delivers the drug, gives mechanical support to the blood vessel and once it is no longer needed the scaffold absorbs into the body leaving no permanent metallic implant.

This same device has been used safely and effectively in the arteries which supply the heart both in clinical trials and current practice and has also been evaluated in the leg arteries in a single-centre pilot study. This study aims to evaluate it's use in a larger number of patients in multiple centres and compare that to a historical control group of metal drug eluting stents. The study will evaluate both ultrasound and angiographic derived patency in those arteries out to a 36 month follow-up time point. This data will be collected in patients who fulfill the inclusion criteria and who are then treated and followed over time.

ELIGIBILITY:
Inclusion Criteria:

* Stenotic (> 50%) or occlusive atherosclerotic disease of the distal popliteal or infrapopliteal arteries
* A maximum of two focal target lesions in one or more distal popliteal or infrapopliteal vessels
* Length of lesion is maximally 55 mm, allowing maximally 2 stents to be implanted
* Reference vessel diameter should be 2.5 mm-4 mm
* Symptomatic critical limb ischemia (Rutherford 3, 4, 5)
* Subject is able to take at least one type of thienopyridine (e.g. clopidogrel) and acetylsalicylic acid
* The patient must be > 18 years of age
* Life-expectancy of more than 12 months
* The patient has no child bearing potential or negative serum pregnancy test within 7 days of the index procedure
* The patient must be willing and able to return to the appropriate follow-up times for the duration of the study
* The patient must provide written patient informed consent that is approved by the ethics committee

Exclusion Criteria:

* Patient refusing treatment
* The reference segment diameter is not suitable for available stent design.
* Unsuccessfully treated (>30% residual stenosis) proximal inflow limiting arterial stenosis
* Untreatable lesion located at the distal outflow arteries
* More than two infrapopliteal lesions in the same limb
* Previously implanted stent(s) or PTA at the same lesion site
* Lesion location requiring kissing stent procedure
* Lesion lies within or adjacent to an aneurysm
* Inflow-limiting arterial lesions left untreated
* The patient has a known allergy to heparin, Aspirin or other anticoagulant/anti-platelet therapies or a bleeding diatheses or is unable, or unwilling, to tolerate such therapies.
* The patient takes Phenprocoumon (Marcumar).
* The patient has a history of prior life-threatening contrast media reaction.
* The patient is currently enrolled in another investigational device or drug trial.
* The patient is currently breast-feeding, pregnant or intends to become pregnant.
* The patient is mentally ill or retarded.
* Subject has received a heart transplant or any other organ transplant or is on a waiting list for any organ transplant
* Subject is receiving or scheduled to receive anticancer therapy for malignancy within 30 days prior to or after the procedure
* Subject is receiving immunosuppression therapy, or has known serious immunosuppressive disease (e.g., human immunodeficiency virus), or has severe autoimmune disease that requires chronic immunosuppressive therapy (e.g., systemic lupus erythematosus, etc.) The patient should also not receive inhibitors of CYP3A (such as Itraconazole, and Erythromycin), or inducers of CYP3A (Cytochrome P450 3A4) (such as Rifampin) within 90 days following the procedure.
* Subject is receiving or is scheduled to receive chronic anticoagulation therapy (e.g., heparin, coumadin)
* Use of alternative therapy (e.g. atherectomy, cutting balloon, laser, radiation therapy) as part of the index procedure

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 4 (Actual)
Dates: Start 2015-06; Primary Completion 2017-06 (Actual); Study Completion 2017-06 (Actual)

PRIMARY OUTCOMES:
Angiographic patency | 12 months
  Freedom from angiographic binary in-scaffold restenosis (>50% stenosis)

SECONDARY OUTCOMES:
Technical success | Procedure
  Technical success defined as the ability to cross and dilate the lesion to achieve residual angiographic stenosis no greater than 30% and residual stenosis less than 50% by duplex ultrasound (US) imaging.
Haemodynamic primary, assisted primary and secondary patency | 1 month
  Haemodynamic primary, assisted primary and secondary patency as assessed by ultrasound
Haemodynamic primary, assisted primary and secondary patency | 6 months
  Haemodynamic primary, assisted primary and secondary patency as assessed by ultrasound
Haemodynamic primary, assisted primary and secondary patency | 12 months
  Haemodynamic primary, assisted primary and secondary patency as assessed by ultrasound
Haemodynamic primary, assisted primary and secondary patency | 24 months
  Haemodynamic primary, assisted primary and secondary patency as assessed by ultrasound
Haemodynamic primary, assisted primary and secondary patency | 36 months
  Haemodynamic primary, assisted primary and secondary patency as assessed by ultrasound
Limb salvage rate (LSR) | 12 months
  Limb salvage defined as 1 minus major amputation rate (major amputation is defined as at or above ankle, as opposed to minor amputation being at or below metatarsus preserving functionality of foot)
Target lesion revascularization (TLR) | 12 months
  Target lesion revascularization (TLR) is defined as a repeat intervention to maintain or re-establish patency within the region of the treated arterial vessel plus 5 mm proximal and distal to the treated lesion edge
Rutherford Category | 12 months
  Clinical success defined as an improvement of Rutherford classification of one class or more as compared to the pre-procedure Rutherford classification
Adverse clinical events | 12 months
  Clinical events defined as fatal, life-threatening, or judged to be severe by the investigator; resulted in persistent or significant disability; necessitated surgical or percutaneous intervention; or required prolonged hospitalization

CONTACTS AND LOCATIONS:
Overall Officials: Ramon L Varcoe, MS,FRACS,PhD, Principal Investigator — Prince of Wales Hospital
Locations (4):
- Australia (2):
  - Prince of Wales Hospital, Sydney, New South Wales
  - Epworth Hospital, Melbourne, Victoria
- Reinier de Graf Hospital, Delft, Netherlands
- Auckland City Hospital, Auckland, New Zealand

IPD SHARING:
Plan to Share IPD: Undecided